CLINICAL TRIAL: NCT03812952
Title: Current Status of Diagnosis and Treatment of Allergic Conjunctivitis in Chinese Ophthalmology Clinic
Brief Title: China Red Eye Study on Allergic Conjunctivitis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiaofeng Lin, associate dean of Zhongshan Ophthalmic Center, Sun Yat-sen University, Sun Yat-sen University
Other Study IDs: Xiaofeng Lin
Record Dates: First submitted 2018-11-08; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Allergic Conjunctivitis
Keywords: misdiagnose; mistreatment; antibiotics
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is the first multi-center cross-sectional study on the diagnosis and misdiagnosis of allergic conjunctivitis in the ophthalmology clinic in China. It provides a clinical basis for the standardized diagnosis and treatment of allergic eye diseases.

DETAILED DESCRIPTION:
Allergic conjunctivitis is a common disease in ophthalmology. The European Allergy Association, Japan, the United States and other countries have clear diagnostic criteria or guidelines for the definition and diagnosis of allergic diseases and allergic conjunctivitis. However, China is currently lacking related guidelines. Allergic conjunctivitis has some of the same symptoms and signs as other infections/non-infectious conjunctival inflammation. When the symptoms and signs are atypical, it is prone to missed diagnosis and misdiagnosis, resulting in prolonged disease duration, drug abuse and waste of medical resources.

The current abuse of antibiotics is considered to be a huge problem in the treatment of ocular surface diseases. A study in our country believes that the rate of misdiagnosis of dry eye is as high as 66.2%, and most of them are misdiagnosed as chronic conjunctivitis, resulting in frequent using a variety of antibiotic eye drops. At present, the misdiagnosis of allergic conjunctivitis and the abuse of antibiotics caused by misdiagnosis in China are still unclear, therefore clinical research is urgently needed. We intend to use this study to understand the status of diagnosis and treatment of allergic conjunctivitis in China, and provide clinical evidence for the standard diagnosis and treatment of allergic eye diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose clinical diagnosis is allergic conjunctivitis.

Exclusion Criteria:

* The investigator believes that there are any unsuitable reasons for participating in the trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients whose clinical diagnosis is allergic conjunctivitis.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Specific diagnosis of the patients | Until the study completion, up to 1 year
  the investigators record the patients' specific diagnosis (such as seasonal allergic conjunctivitis, perennial allergic conjunctivitis, vernal keratoconjunctivitis，and etc) on questionnaire when the patient come

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Lin, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center of Sun yat-sen Universtiy, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No